CLINICAL TRIAL: NCT03947047
Title: Detection of Placenta Accreta by Means of Volatile Organic Compounds in Exhaled Women Breath. A Prospective Case Control Study.
Brief Title: Detection of Placenta Accreta Via Exhaled Women Breath
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Collaborators: Technion, Israel Institute of Technology (Other)
Responsible Party: Principal Investigator, Sivan Easton, Principal Investigator, HaEmek Medical Center, Israel
Other Study IDs: 0021-19-EMC
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Placenta Accreta, Third Trimester
Keywords: Exhaled Women Breath; Placenta Accreta; Ultrasound
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Organic Compounds in Exhaled Women Breath and blood samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Placenta Accreta: Women found to have abnormal placentation (any degree of placenta accreta) during the cesarean section.
  Interventions: Diagnostic Test: NA-NOSE
- No Placenta Accreta: Women found to have normal placenta separation during the cesarean section.
  Interventions: Diagnostic Test: NA-NOSE

INTERVENTIONS:
Diagnostic Test: NA-NOSE — Breath and blood samples for distinguishing biomarkers.

SUMMARY:
Placenta accreta is a relatively rare event, in which the placenta is abnormally implanted into the uterine myometrium. The most significant complication is intense bleeding, mainly during labor. The incidence of placenta accreta increased during the last years due to the increase in cesarean delivery rate, which is the main risk factor. Pre-cesarean diagnosis of placenta accreta may improve surgical outcome. Early diagnosis allows appropriate preparation of multidisciplinary team (including, among others; OB-GYN, urologists, anesthesiologists, neonatologists) and massive blood products. Pre-cesarean diagnosis is based on imaging, mainly ultra-sound. This modality has significant false positive rate which may result in extreme sources investment and even indicated pre-term labor, in vain. Volatolome is a complex of volatile markers emitted in several processes in the human body and collected from breath, skin, urine, blood, feces and more. This profile may be used to identify volatile markers for specific medical conditions. NA-NOSE is an electronic device knowing to identify differences in the Volatolome between "healthy" and "sick" subjects. The objective of this study is to identify specific volatile profile for placenta accreta which will help to distinguish between women with placenta accreta and those without.

DETAILED DESCRIPTION:
Pregnant women with clinical risk factors for placenta accreta will perform targeted sonographic evaluation for detection of placenta accreta features, according to a standard protocol. Of those with clinical and sonographic risk factors who will agree to participate in the study, will be asked to breathe through a collection device (NA-NOSE) for "lung wash". The participant will be instructed to inhale through the device and exhale to the ambient air for about 3 minutes. After the lung wash step, the collector will inform the participant that she is about to start filling the collective bags. At the end of a regular breath, after exhaling, the collector will ask the participant to take a deep breath so the full volume of the lungs is filled, and then exhale until both the dead space bag and collection bag are full. After filling the first bag, a second bag will be placed and the participant will be asked to repeat the act. In addition, a venous blood sample of 8-10 ml will be taken from each participant.

The samples will be transferred to the Department of Chemical Engineering and Russell Berrie Nanotechnology Institute, Technion-Israel, Institute of Technology. The samples will be analyzed to determine the nature and composition of the volatile biomarkers in the related breath and blood samples.

In this way, the investigators will identify among women who have clinical and sonographic risk factors for placenta accreta, those biomarkers distinguishing women with placenta accreta (group 1) from those who will not have placenta accreta at birth (group 2).

ELIGIBILITY:
Inclusion Criteria:

1. Pregnancy > 28 weeks of gestation.
2. Agreement to participate and sign an informed consent.
3. Ability to give breath and blood samples.
4. Risk factors for placenta accreta:

   1. Placenta previa.
   2. Previous 1 or more cesarean sections with placenta in the scar area.
   3. Previous uterine procedures (myomectomy, curretage) and sonographic suspicion of abnormal placentation.

      - Exclusion Criteria: None

      -

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women, 28 weeks of gestation or more, with known risk factors for placenta accreta referred to our institute to perform an ultrasound scan for detecting abnormal placentation.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-08-06 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Detection of placenta accreta | 2 years
  The aim of the study is to improve pre-cesarean detection of placenta accreta using volatile biomarkers appearing in exhaled breath and/or blood samples, using a simple inexpensive tool termed NA-NOSE.

CONTACTS AND LOCATIONS:
Overall Officials: Sivan Easton, MD, Principal Investigator — Emek Medical Center
Locations (1):
- HaEmek Medical Center, Afula, Israel

IPD SHARING:
Plan to Share IPD: Undecided
Decision regarding IPD sharing, will be taken later.